CLINICAL TRIAL: NCT00282139
Title: Aripiprazole in the Treatment of Tourette's Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSARIP703 / WIRB #20031378; 00040256/00042966
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Tourette's Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
This is an open-label, flexible dose study designed to evaluate the safety and efficacy of aripiprazole in TS (or chronic tic disorder) subjects with or without associated OC symptoms and with or without ADHD symptoms.

DETAILED DESCRIPTION:
This is an open-label, flexible dose study designed to evaluate the safety and efficacy of aripiprazole in TS (or chronic tic disorder) subjects with or without associated OC symptoms and with or without ADHD symptoms.

ELIGIBILITY:
Inclusion Criteria:

DSM-IV primary diagnosis of Tourette's syndrome or chronic tic disorder;

"Moderate" severity as reflected on the CGI or the YGTSS;

Normal ECG; and,

Written informed consent/assent.

Exclusion Criteria:

Female subjects of childbearing potential who are not practicing an effective method of birth control (including abstinence);

Subjects who are pregnant or nursing women;

Subjects with known seizure disorder, a history or seizures or with conditions that lower seizure threshold;

Subjects who currently meet DSM-IV criteria for: Schizophrenia, Schizoaffective Disorder, Delusional Disorder, or Psychotic Disorder Not Otherwise Specified;

Subjects with a Psychoactive Substance Abuse disorder (within the past 3 months);

Subjects with known allergy or hypersensitivity to aripiprazole;

Subjects who have any depot neuroleptic within one treatment cycle or any other changes in psychoactive medications (with the exception of antidepressants) in one month and two months for antidepressants prior to study entry for first administration of study medication;

Subjects who have clinically significant abnormalities based on physical examination, medical history, ECG, or laboratory tests; and,

Subjects on medication that pose drug interaction potential with aripiprazole such as carbamazepine, ketoconazole, paroxetine, and fluoxetine.

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2004-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Global improvement in severity of symptoms (tic behaviors)

SECONDARY OUTCOMES:
Assessment of behavior (improvement and severity) for co-morbid conditions, OCD and/or ADHD

CONTACTS AND LOCATIONS:
Overall Officials: Tanya K Murphy, M.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States